CLINICAL TRIAL: NCT04010760
Title: Non-invasive Diagnosis of Pulmonary Embolism by Use of Biomarkers in Exhaled Breath Condensate
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Inger Lise Gade, MD, PhD, Registrar, Aalborg University Hospital
Other Study IDs: ILG-PE-2018; #0053310 (Other Grant/Funding Number: The Novo Nordisk Foundation); N-20180086 (Other: Den Videnskabsetiske Komite for Region Nordjylland)
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. Exhaled breath condensate (EBC)
  2. Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PE confirmed: Patients admitted with confirmed pulmonary embolism.
  Interventions: Diagnostic Test: Test of biomarkers for PE in EBC
- PE suspected: Patients admitted with suspected, but not confirmed pulmonary embolism.
  Interventions: Diagnostic Test: Test of biomarkers for PE in EBC
- Controls: Healthy controls same gender and age (within af range of 10 years) as PE patients
  Interventions: Diagnostic Test: Test of biomarkers for PE in EBC

INTERVENTIONS:
Diagnostic Test: Test of biomarkers for PE in EBC — New method for diagnosis of pulmonary embolism (PE) in order to validate/consolidate 151 putative identified biomarkers for PE in the exhaled breath condensate (EBC).
  The EBC will be collected by use of the RTube(R) system which has been used in previous studies of EBC. As the patient breathes through a mouth piece, the exhaled breath is led through a cooling chamber where the vaporous part of the exhaled breath condenses.
  We aim at collecting a total minimum of 3.0 mL EBC per study subject in order to have a sufficient amount of protein for the subsequent analysis. We aim at collecting exhaled breath condensate for 2*15 minutes with the possibility to stop the collection after less than 15 minutes if the volume is sufficient.

SUMMARY:
In this study, a new, non-invasive method for diagnosis of pulmonary embolism (PE) will be tested. In pre-clinical studies, we have identified 151 putative biomarkers for pulmonary embolism in the exhaled breath condensate (EBC). These biomarkers needs validation/consolidation in a clinical setting before further test of this new diagnostic method.

DETAILED DESCRIPTION:
The study will compare the protein profiles of EBC collected from patients admitted to the department of cardiology with suspected pulmonary embolism and controls with same age (within a range of 10 years) and gender from the outpatient clinic awaiting elective cardiovascular surgery. The main-outcome (i.e. means of the relative amounts of specific proteins in the EBC samples) will be compared by unpaired t-tests after assessment of normality and standard deviations within the three groups (PE confirmed, PE suspected but not confirmed and controls). Furthermore, sensitivity and specificity will be calculated for relevant proteins. The results from analysis of EBC samples from the patients and controls will be compared with results from the porcine model in order to confirm and reduce the number of putative biomarkers for PE. Blood samples (i.e. excess plasma from routine blood samples drawn as a part of routine diagnostic work-up) from the study participants will be stored for standardization of the putative markers and verification and supplementing analysis of the EBC markers. In order to qualify the most suitable markers and substrates for standardization, the analysis of the EBC samples must be completed before the blood samples can be analyzed. Only biochemical, no genetic analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria - Suspected/confirmed PE patients:

* Admitted to the emergency department with initial diagnosis of PE, visited to the Department of Cardiology at Aalborg University Hospital.
* Are conscious and able to understand the given study information.
* Possess legal capacity.
* Age above 18 years.
* Informed, signed consent is obtained.
* Clinically stable, which is defined as patients with stable blood pressure and not in need for other treatments .
* No need for organ support, which comprises need for vasopressors or inotropes, mechanical ventilation, extra corporal circulation or renal replacement therapy.

Inclusion Criteria - Controls:

• Patients as the PE patients, but where the diagnosis of PE is rejected.

The rest of the control persons will be recruited as described:

* Patients who are going to have elective procedures at the Department of Cardiology, Aalborg University Hospital.
* Same gender and age (within a 10-year range) as an included PE patient.
* Are conscious and able to understand the given study information.
* Possess legal capacity.
* Age above 18 years.
* Informed, signed consent is obtained.

Exclusion Criteria:

* Active malignant disease (i.e. ongoing anti-cancer therapy or palliation).
* Current smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is expected that
  * 40 patients with confirmed PE,
  * 40 patients with suspected PE, but where diagnostic work-up did not confirm PE and
  * 40 healthy controls
  will be included in the study over a six-month period.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Prediction of pulmonary embolism by use of biomarkers in the EBC | 1-2 years
  The primary outcome is prediction of pulmonary embolism by use of one or more novel biomarkers in the EBC.

CONTACTS AND LOCATIONS:
Overall Officials: Inger L Gade, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gade IL, Riddersholm SJ, Stilling-Vinther T, Brondum RF, Bennike TB, Honore B. A clinical proteomics study of exhaled breath condensate and biomarkers for pulmonary embolism. J Breath Res. 2023 Nov 17;18(1). doi: 10.1088/1752-7163/ad0aaa. PMID 37939397